CLINICAL TRIAL: NCT03520530
Title: Mouth Guard Use in the Second Stage of Labor: A Randomized Controlled Trial
Brief Title: Mouth Guard Use in the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 37133
Record Dates: First submitted 2018-03-23; First posted 2018-05-09 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Dystocia; Fetal; Labor Long; Cesarean Section, Affecting Fetus or Newborn
Keywords: second stage; spontaneous vaginal delivery
MeSH Terms: conditions — Dystocia | interventions — Mouth Protectors

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial in which patients who make it to the second stage of labor will be randomized to wear a mouth guard while pushing during the second stage of labor or continue through the second stage of labor without a mouth guard. They will be randomized in a 1:1 fashion using RedCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mouth Guard (Experimental): Patients will push in the second stage of labor without use of mouth guard
  Interventions: Device: Mouth Guard
- Control (No Intervention): Patients will push in the second stage of labor without use of mouth guard

INTERVENTIONS:
Device: Mouth Guard — Patient will wear mouth guard while pushing in the second stage of labor
  Arms: Mouth Guard

SUMMARY:
Shortening the second stage of labor, the time spent pushing the baby out, is important for positive mother and infant's outcomes. Lack of progress of labor for any reason is the most common reason for cesarean section in women having their first baby and the second most common reason for cesarean section in women who have already had a baby. In 2014, a large study done across the United States showed increases in complications in both mother and infant when pushing was prolonged, including uterine infection, postpartum hemorrhage, more extensive vaginal tearing, shoulder dystocia, 5 minute Apgar score less than 4, infant admission to Neonatal Intensive Care Unit and neonatal infections. Therefore, the challenge is to consider alternative practices in order to maximize a mother's chance of a vaginal delivery and minimize these associated risks to both mother and baby.

Mouth guards are used primarily in contact sports, and have been demonstrated to reduce or prevent injury to the teeth. Additionally, it has been proposed that wearing a mouth guard increases the strength of different muscle groups. A recent randomized controlled pilot study including women with their first pregnancy using a dental support device (DSD) during the second stage of labor evaluated the length of the second stage and outcomes. They found a significant decrease of 38% in the length of pushing time in the group that used a DSD. Additionally, there was a decreased rate of cesarean section in this group, however a p-value was not reported. This study only included 64 patients. A second, larger trial did not find a significant difference in pushing time, however the rate of interventions such as a vacuum or forceps-assisted vaginal delivery and cesarean section were much higher in the control group due to prolonged pushing. The results of the second study are contradictory in nature, yet the researchers do not provide hypotheses into why this may be.

It is clear from the previously mentioned studies that further research is needed. Our hypothesis is that using such a device would help women to push more effectively during the second stage of labor thus shortening the time needed to push the baby out and increasing the rate of vaginal delivery. The purpose of this study is to determine whether wearing a mouth guard in the second stage of labor affects the length of the second stage of labor and improves mother & infant outcomes.

DETAILED DESCRIPTION:
Optimizing the second stage of labor is important for positive maternal and neonatal outcomes. Dystocia of labor refers to a lack of progress of labor for any reason, and it is the most common indication for cesarean delivery in nulliparous women and the second most common indication for cesarean delivery in multiparous women. In 2014, a large US multicenter cohort study showed increases in maternal and neonatal morbidities when the second stage was prolonged, including chorioamnionitis, postpartum hemorrhage, 3rd and 4th degree perineal laceration, shoulder dystocia, 5 minute Apgar score less than 4, neonatal admission to NICU and neonatal sepsis. Therefore, clinicians are challenged to consider alternative practices in order to maximize a mother's chance of a normal delivery and minimize these associated risks to both mother and baby.

Mouth guards are used primarily in contact sports, and have been demonstrated to reduce or prevent injury to the teeth. Most commonly made of synthetic polymers, mouth guards function as a shock-absorber. Even among sports medicine literature, there is a call for more research into use and education about protective gear. Previous studies have shown that wearing a mouth guard increases the isometric strength of different muscle groups. Recent studies have begun to explore whether wearing a similar style mouth guard will shorten the duration of the second stage of labor. A recent randomized controlled pilot study including nulliparous women using a dental support device (DSD) during the second stage evaluated the length of the second stage and outcome thereof. They defined the second stage of labor as the time between complete cervical dilation and fetal expulsion. They found a significant decrease of 38% in the length of the second stage in the group that used a DSD. Additionally, there was a decreased rate of cesarean section in this group, however a p-value was not reported. This study only included 64 patients. A second, larger trial also looking at nulliparous women did not find a significant difference in length of second stage of labor however the rate of obstetrical interventions such as operative vaginal delivery and cesarean section were much higher in the control group due to prolonged second stage of labor. Though the results of the second study are contradictory in nature, the researchers do not provide hypotheses into why this may be.

Our hypothesis is that using such a device would help women to push more effectively during the second stage of labor thus shortening the second stage and increasing the rate of spontaneous vaginal deliveries that do not require operative intervention. Developing a way to shorten the second stage of labor and reduce the number of cesarean sections or instrumental deliveries could reduce the morbidity of mothers and their infants and decrease health care spending.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Age 18-55
* Presenting for delivery at Christiana Care Health Services
* Singleton pregnancy
* Cephalic pregnancy
* Term pregnancy

Exclusion Criteria:

* Multiple gestation
* Known uterine anomalies, excluding resected uterine septums and fibroids
* Estimated fetal weight less than 10th% for gestation age with abnormal umbilical dopplers
* Estimated fetal weight less than the 5th percentile
* History of cardiac disease requiring assisted second stage of labor
* Oral implants, braces or active dental infection precluding mouth guard use
* Preeclampsia with severe features treated with magnesium sulfate
* History of shoulder dystocia
* History of myomectomy
* Maternal history of myasthenia gravis
* Maternal history of sleep apnea with home CPAP use
* Category III fetal heart tracing
* Active vaginal bleeding consistent with placental abruption
* Diagnosis of chorioamnionitis prior to start of second stage of labor
* Participation in another interventional research study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Time of Second Stage of Labor | Time from full cervical dilation (10cm) to delivery of the fetal head, approximately 2 hours
  Time in minutes

SECONDARY OUTCOMES:
Mode of Delivery | From time of randomization until delivery, up to one week
  Spontaneous vaginal delivery, assisted vaginal delivery, cesarean section
Instrumental Delivery | From time of randomization until delivery, up to one week
  Type of instrument used in assisting delivery
Patient Satisfaction | From time of randomization until delivery, up to one week
  Patient satisfaction with device as measured by survey
Perineal Laceration | From time of randomization until delivery, up to one week
  Degree of perineal laceration with vaginal delivery
Apgar Score | From 0 to 10 minutes after delivery
  Apgar scores of infants at 1, 5, and 10 minutes
Percentage of Time Spent Using Device | From time of randomization until delivery, up to one week
  Provider will estimate percentage of second stage that patient used device
Neonatal ICU Admission Rate | From time of randomization until delivery, up to one week
  Number of infants admitted to the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shy, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to submit for publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year

REFERENCES:
- [Background] Gabbe, Steven G., Jennifer R. Niebyl, Joe Leigh Simpson, and Garland D. Anderson. 1991. Obstetrics: normal and problem pregnancies. New York: Churchill Livingstone.
- [Background] Laughon SK, Berghella V, Reddy UM, Sundaram R, Lu Z, Hoffman MK. Neonatal and maternal outcomes with prolonged second stage of labor. Obstet Gynecol. 2014 Jul;124(1):57-67. doi: 10.1097/AOG.0000000000000278. PMID 24901265
- [Background] Vidovic-Stesevic V, Verna C, Krastl G, Kuhl S, Filippi A. Facial and Dental Injuries in Karate. Swiss Dent J. 2015;125(7-8):810-4. doi: 10.61872/sdj-2015-07-08-01. PMID 26345152
- [Background] Farrington T, Onambele-Pearson G, Taylor RL, Earl P, Winwood K. A review of facial protective equipment use in sport and the impact on injury incidence. Br J Oral Maxillofac Surg. 2012 Apr;50(3):233-8. doi: 10.1016/j.bjoms.2010.11.020. Epub 2011 Feb 3. PMID 21295384
- [Background] Arent, S., McKenna, J. and Golem, D. (2010). Effects of a neuromuscular dentistry-designed mouthguard on muscular endurance and anaerobic power. Comparative Exercise Physiology, 7(02), pp.73-79.
- [Background] Matsuo K, Mudd JV, Kopelman JN, Atlas RO. Duration of the second stage of labor while wearing a dental support device: a pilot study. J Obstet Gynaecol Res. 2009 Aug;35(4):672-8. doi: 10.1111/j.1447-0756.2008.01010.x. PMID 19751326
- [Background] Aviram A, Ashwal E, Hiersch L, Hadar E, Wiznitzer A, Yogev Y. The effect of intrapartum dental support use among nulliparous during the second stage of labor - a randomized controlled study. J Matern Fetal Neonatal Med. 2016 Mar;29(6):868-71. doi: 10.3109/14767058.2015.1024648. Epub 2015 Mar 19. PMID 25777794